CLINICAL TRIAL: NCT03019991
Title: A Study on Safety, Tolerability and Pharmacokinetics of Ritonavir-boosted Danoprevir in Single and Multiple Doses in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Danoprevir/r in Healthy Volunteers China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASC08201501
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: pharmacokinetics,Danoprevir
MeSH Terms: interventions — danoprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PK Group (Danoprevir,Ritonavir) (Experimental): Danoprevir(DNV)administered orally 100mg QD on day 1, day 4 and day 14;100mg BID on day 5 -day 13; Ritonavir administered orally 100mg QD on day 4 and day 14; 100mg BID on day 5 -day 13;
  Interventions: Drug: Danoprevir; Drug: Ritonavir
- Placebo Group (Placebo Comparator): ASC 08 Placebo administered orally 100mg QD on day 1, day 4 and day 14; 100mg BID on day 5 -day 13; Ritonavir administered orally 100mg QD on day 4 and day 14; 100mg BID on day 5 -day 13 for 14 days;
  Interventions: Drug: Ritonavir; Drug: Placebo

INTERVENTIONS:
Drug: Danoprevir — Danoprevir(DNV)administered orally 100mg QD on day 1, day 4 and day 14; 100mg BID on day 5 -day 13
  Other Names: ASC08
  Arms: PK Group (Danoprevir,Ritonavir)
Drug: Ritonavir — Ritonavir administered orally 100mg QD on day 4 and day 14; 100mg BID on day 5 -day 13
  Other Names: RTV
Drug: Placebo — ASC 08 Placebo administered orally 100mg QD on day 1, day 4 and day 14; 100mg BID on day 5 -day 13
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics of Danoprevir in single dose (100mg QD on day 1, day 4 and day 14) and Ritonavir-boosted Danoprevir (100mg QD on day 4 and day 14) in single and multiple doses (100mg BID on day 5 -day 13) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Healthy men or women based on history, physical examination, laboratory examination and ECG.
* Negative serum or urine pregnancy test result (sensitivity of 25 mIU or better) for women with childbearing potential within the 24-hour period before the first dose of study drugs
* Female patients with childbearing potential (menopause within 1 year) must agree to use two reliable forms of effective non-hormonal contraception (i.e., condoms, cervical barriers, intrauterine device, spermicides, or sponge), at least 1 of which must be a physical barrier method, during treatment and for at least 6 months following the last dose of ribavirin
* All male patients with female partners of childbearing potential must use two reliable forms of effective contraception (combined) during treatment and for 6 months following the last dose of ribavirin
* Others as specified in the detailed protocol

Exclusion Criteria:

* Have medical history, or has disease, such as cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, blood system, nerve system disease or psychiatric disease and acute or chronic infectious diseases and malignant tumors.
* Has a history of drug or food allergy.
* Positive hepatitis A antibody，positive hepatitis B surface antigen， positive hepatitis C antibody，syphilis antibody or HIV antibody at screening.
* Had gastrointestinal surgery, vagotomy, intestinal resection or any possible interference with gastrointestinal peristalsis, pH or absorbed by surgery.
* Pregnant, lactating or menstrual period and unwilling to reliable contraception period women of childbearing age.
* Female partners have fertility and reliable contraceptive measures of men.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 40 days
Pharmacokinetics: Maximum plasma concentration at steady-state (Css,max) | Up to 16 days
Pharmacokinetics: Total area under the concentration-time curve form time 0 to 12 hours post-dose at steady-state | Up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Huoling Tang, PhD, Study Director — Ascletis Pharmaceuticals Co., Ltd.

IPD SHARING:
Plan to Share IPD: No